CLINICAL TRIAL: NCT02543138
Title: The Development and Experimental Application of a New Thoracostomy Trocar
Acronym: TDEANTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Clinical Fellow, Hanyang University
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: LEE YOON-JE
Record Dates: First submitted 2015-08-14; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed thoracostomy (Experimental): Closed thoracostomy using the new trocar by novice
  Interventions: Device: Trocar

INTERVENTIONS:
Device: Trocar — Closed thoracostomy using the new trocar

SUMMARY:
Traditional closed thoracostomy exhibit certain shortcomings. Blind dissection is a lengthy process that is difficult for unskilled physicians, whereas the use of a traditional trocar is relatively likely to damage internal organs. In this study, investigators developed a new trocar and examined its usefulness.

DETAILED DESCRIPTION:
The new trocar consists of a mold and a stylet; the mold has a hole in its side to ensure that the chest tube proceeds in only one direction. The mold also has a mark to indicate insertion depth. Sixteen participants without experience with thoracostomies observed one closed thoracostomy procedure using the new trocar and then performed three thoracostomies on a cadaver. For each of these thoracostomies, investigators measured the time required for chest tube insertion, the position of the tip of the chest tube within the thoracic cavity, the difficulty associated with the procedure, and the volunteer's confidence after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Senior medical students without prior experience with closed thoracostomies

Exclusion Criteria:

* Wrist disease, Pregnancy, Do not want to participate

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time to closed thoracostomy | 5 minutes

SECONDARY OUTCOMES:
The accuracy of the position of the tip of the chest tube | 5 minutes
  Yes or No

OTHER OUTCOMES:
Scale of procedural difficulty | within 2 minutes
  Score range from 0[Easy] to 10 [Difficult]
Scale of procedural confidence | within 2 minutes
  Score range from 0 [confidence : no] to 10 [confidence : yes]

CONTACTS AND LOCATIONS:
Overall Officials: YOON-JE LEE, Master, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University, College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lee YJ, Choi HJ, Lim TH, Lee SH, Hwang SJ. The development and experimental application of a new thoracostomy trocar. Am J Emerg Med. 2016 May;34(5):917-20. doi: 10.1016/j.ajem.2016.02.016. Epub 2016 Feb 12. No abstract available. PMID 26964824